CLINICAL TRIAL: NCT00405574
Title: A Randomized, Phase II Study of Two Dose Levels of ATN-224 in Patients With Biochemically Relapsed, Early Stage Prostate Cancer Not on Hormone Therapy
Brief Title: Study of ATN-224 in Patients With Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Attenuon (Industry)
Collaborators: Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Jennifer Callahan, Senior Manager, Clinical Development, Attenuon, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN-224-005
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Prostate Cancer
Keywords: prostate; PSA; antiangiogenic; copper; ATN-224
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tetrathiomolybdate

ARMS (2):
- High Dose (Experimental): ATN-224 dose 300mg
  Interventions: Drug: ATN-224
- Low Dose (Experimental): ATN-224 dose: 30mg
  Interventions: Drug: ATN-224

INTERVENTIONS:
Drug: ATN-224 — ATN-224 high dose: 300mg ATN-224 low dose: 30mg

SUMMARY:
This is a multicenter, randomized, phase II study of the safety and efficacy of two dose levels of oral ATN-224 in patients with prostate cancer with a rising serum PSA in the absence of detectable disease. Patients will be randomized (1:1) after confirmation of eligibility requirements. The primary endpoint is to determine the proportion of patients who do not have PSA progression for 24 weeks. PSA progression is defined as at least a 50% increase in PSA and >5 ng/mL from baseline or post-treatment nadir if lower than baseline, confirmed by another PSA at least 28 days later.

DETAILED DESCRIPTION:
ATN-224 is an orally active, small molecule that has been shown in cellular and animal models to be anti-angiogenic and to have activity against prostate cancer cell lines. ATN-224 has the potential to affect the progression of prostate cancer by mechanisms that include both antiangiogenic and antitumor pathways. ATN-224 may change the time to overt metastatic disease in patients with rising PSA as the only manifestation of disease after treatment with curative intent and delay the need for hormonal therapies.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically confirmed, localized prostate cancer who have a prostate-specific antigen (PSA) doubling time (DT) as calculated according to the Memorial Sloan-Kettering Cancer Center nomogram (http://www.mskcc.org/mskcc/html/10088.cfm)

  * Doubling time < 12 months after local therapy in patients who have not had any previous hormone therapy, or
  * Doubling time < 12 months starting at least 6 months after their last dose of hormone therapy
* Patients must have a serum testosterone >150 ng/dL at the time of study entry. Patients may have received previous castrating hormonal therapy or anti-androgens, provided that the testosterone level is >150 ng/dL at the time of study entry. Prior chemotherapy is also allowed as long as the requirements for adequate organ and marrow function are met.
* No detectable disease as assessed by physical examination and bone and CT (abdomen and pelvis) scans within 4 weeks prior to the first dose of ATN-224
* A minimum of three PSA values, each at least 4 weeks apart, to calculate PSA-DT. The last PSA level prior to enrollment must be at least 2.0 ng/mL and be rising over the prior value.
* Age ≥18 years
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥50%; see Appendix A)
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/uL
  * platelets ≥100,000/uL
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤2 X institutional upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤2 X ULN
  * creatinine clearance (measured or calculated) ≥30 mL/min
  * serum testosterone >150 ng/mL or return to pre-treatment values for patients who received hormone therapy

Patients are allowed to receive erythropoietin or blood transfusions before receiving their first dose of ATN-224 to bring the hemoglobin level to >9 g/dL to meet eligibility criteria.

* At least 28 days from receiving any investigational agent
* The effects of ATN-224 on sperm at the recommended therapeutic dose are unknown. For this reason men with partners of child-bearing potential must agree to use adequate contraception (hormonal and/or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation through the follow up visit 28 days after the last dose of ATN-224
* Willingness to forgo taking copper- or zinc-containing vitamins or supplements
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* Patients who have had radiotherapy within 3 months prior to the first dose of ATN 224
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ATN-224 or omeprazole or other long acting antacids
* History of malabsorption syndromes or other gastrointestinal disorders that may affect ATN-224 absorption, including bowel obstruction, celiac disease, sprue, cystic fibrosis
* Ineligible to receive either omeprazole (Prilosec®), lansoprazole (Prevacid®), pantoprazole (Protonix®), or ranitidine (Zantac®)
* Inability to swallow study medication capsules
* Other serious medical or psychiatric illness preventing informed consent or with the potential to interfere with assessment of safety or efficacy of ATN-224 treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients known to be positive for HIV or infectious hepatitis type A, B or C
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer or any other cancer from which the patient has been disease-free for 5 years
* Patients receiving steroid therapy for concurrent illness unless they have been on a stable dose for 3 months.
* Patients receiving hormonal therapy including gonadotropin-releasing hormone agonist/antagonist, antiandrogens, diethylstilbestrol, any other estrogen-like agents, any hormonally active over-the-counter compounds such as PC-SPES or finasteride

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-06 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Determine the proportion of patients who have not had prostate specific antigen (PSA) progression for 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Establish the safety of the two dose levels of ATN-224 | Ongoing
Determine the proportion of patients with a 50% reduction from baseline of PSA confirmed by a second PSA value at least 28 days later | End of Study
Determine the change in PSA doubling time (PSA-DT) from baseline | End of Study
Determine the maximal % decrease in PSA after treatment | End of Study
Determine the time to PSA progression (as defined by this protocol) | End of Study
Determine the 24-week rate of metastases | 24 weeks
Determine the effect of ATN-224 treatment on levels of Cu,Zn-superoxide dismutase (SOD1) in red blood cells | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gordon, MD, Study Director
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin